CLINICAL TRIAL: NCT02875808
Title: Early Detection of CSF Infection in Neurosurgical Patients
Brief Title: Cerebrospinal Fluid IL-6, IL-8 and PCT as Early Marker of an Intrathecal Infection in Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Sascha Marx, Dr. med., University Medicine Greifswald
Other Study IDs: CSF IL-6, IL-8 and PCT
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Intrathecal Infection; External Ventricular Drainage Associated Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients: patients with an external ventricular drainage

SUMMARY:
The value of CSF IL-6, IL-8 and Procalcitonin in detecting an early diagnosis of intrathecal infection in neurosurgical patients with an external ventricular drainage is evaluated.

DETAILED DESCRIPTION:
The value of CSF IL-6, IL-8 and Procalcitonin in detecting an early diagnosis of intrathecal infection in neurosurgical patients with an external ventricular drainage is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* external ventricular drainage
* informed consent

Exclusion Criteria:

* no informed consent
* prior intrathecal infection
* prior systemic infection / sepsis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients with an external ventricular drainage
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
increasing IL-6, IL-8 and PCT prior to an clinically apparent intrathecal infection/ a detection with the goldstandard | 08/ 2014 - 12/ 2016

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided